CLINICAL TRIAL: NCT02746809
Title: Medtronic CoreValve Evolut R United States Clinical Study (Evolut 34R Addendum)
Brief Title: Medtronic CoreValve Evolut R U.S. Clinical Study (Evolut 34R Addendum)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10211838DOC
Record Dates: First submitted 2016-04-18; First posted 2016-04-21 (Estimated); Results first posted 2017-12-29 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CoreValve Evolut 34R TAVR system (Experimental): Treatment of Aortic Stenosis with Medtronic CoreValve Evolut R 34R TAVR System.
  Interventions: Device: CoreValve Evolut 34R TAVR system

INTERVENTIONS:
Device: CoreValve Evolut 34R TAVR system — The CoreValve Evolut 34R System is a transcatheter aortic valve implantation system comprised of the following three components:
  1. Evolut 34R Transcatheter Aortic Valve (TAV)
  2. EnVeo R Delivery Catheter System (DCS) with EnVeo R InLine Sheath
  3. EnVeo R Loading System (LS)

SUMMARY:
The study objectives are to assess the safety and efficacy of the CoreValve Evolut 34R transcatheter aortic valve replacement (TAVR) system in patients with severe symptomatic aortic stenosis who are considered at high or extreme risk for surgical aortic valve replacement.

DETAILED DESCRIPTION:
This objective will be accomplished by a prospective, single arm, historical controlled, multi-site study involving up to 60 implanted subjects at up to 15 study sites in the United States. Procedural and 30 day safety and efficacy results from this study will be compared to appropriate historical control data for the Medtronic CoreValve System. Subjects will be followed up to 5 years following implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Severe aortic stenosis, defined as aortic valve area of < 1.0 cm2 (or aortic valve area index of < 0.6 cm2/m2) by the continuity equation, AND mean gradient > 40 mmHg or maximal aortic valve velocity > 4.0 m/sec by resting echocardiogram.

   Subjects with low-flow/low gradient severe aortic stenosis can be included, provided low-dose dobutamine or exercise stress echocardiography demonstrates a mean gradient of > 40 mmHg or a maximal aortic valve velocity of > 4.0 m/sec, AND aortic valve area of < 1.0 cm2 (or aortic valve area index of < 0.6 cm2/m2).
2. Society of Thoracic Surgeons (STS) score of ≥ 8 OR documented heart team agreement of ≥ high risk for aortic valve replacement due to frailty or co-morbidities.
3. Symptoms of aortic stenosis, AND New York Heart Association (NYHA) Functional Class II or greater.
4. The subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits.

   Exclusion Criteria:
5. Any condition considered a contraindication for placement of a bioprosthetic valve (e.g. subject is indicated for mechanical prosthetic valve).
6. A known hypersensitivity or contraindication to any of the following which cannot be adequately pre-medicated:

   * aspirin or heparin (HIT/HITTS) and bivalirudin
   * ticlopidine and clopidogrel
   * Nitinol (titanium or nickel)
   * contrast media
7. Blood dyscrasias as defined: leukopenia (WBC < 1000 mm3), thrombocytopenia (platelet count <50,000 cells/mm3), history of bleeding diathesis or coagulopathy, or hypercoagulable states.
8. Untreated clinically significant coronary artery disease requiring revascularization.
9. Severe left ventricular dysfunction with left ventricular ejection fraction (LVEF) < 20% by echocardiography, contrast ventriculography, or radionuclide ventriculography.
10. End stage renal disease requiring chronic dialysis or creatinine clearance < 20 cc/min.
11. Ongoing sepsis, including active endocarditis.
12. Any percutaneous coronary or peripheral interventional procedure with a bare metal or drug eluting stent performed within 30 days prior to study procedure.
13. Symptomatic carotid or vertebral artery disease or successful treatment of carotid stenosis within 10 weeks of Heart Team assessment.
14. Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or mechanical hemodynamic support.
15. Recent (within 6 months of Heart Team assessment) cerebrovascular accident (CVA) or transient ischemic attack (TIA).
16. Gastrointestinal (GI) bleeding that would preclude anticoagulation.
17. Subject refuses a blood transfusion.
18. Severe dementia (resulting in either inability to provide informed consent for the study/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits).
19. Estimated life expectancy of less than 12 months due to associated non-cardiac co-morbid conditions.
20. Other medical, social, or psychological conditions that in the opinion of the investigator precludes the subject from appropriate consent or adherence to the protocol required follow-ups exams.
21. Currently participating in an investigational drug or another device study (excluding registries).
22. Evidence of an acute myocardial infarction ≤ 30 days before the study procedure.
23. Need for emergency surgery for any reason.
24. Liver failure (Child-Pugh class C).
25. Subject is pregnant or breast feeding.

    Anatomical exclusion criteria:
26. Pre-existing prosthetic heart valve in any position.
27. Mixed aortic valve disease (aortic stenosis with severe aortic regurgitation).
28. Severe mitral regurgitation.
29. Severe tricuspid regurgitation.
30. Moderate or severe mitral stenosis.
31. Hypertrophic obstructive cardiomyopathy.
32. Echocardiographic or Multi-Slice Computed Tomography (MSCT) evidence of intracardiac mass, thrombus, or vegetation.
33. Congenital bicuspid or unicuspid valve verified by echocardiography.

    For transfemoral or transaxillary (subclavian) access:
34. Access vessel diameter < 5.5 mm or <6.0 mm for patent left internal mammary artery (LIMA)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-06; Primary Completion 2016-11 (Actual); Study Completion 2021-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathew R Williams, MD, Principal Investigator — NYU Langone Medical Center
Locations (10):
- United States (10):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - New York Langone Medical Center, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Riverside Methodist Hospital, Columbus, Ohio
  - Pinnacle Health/Moffitt Heart and Vascular Institute, Harrisburg, Pennsylvania
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Aurora Health Care/St Luke's Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- CoreValve Evolut R TAVR System 34R Valve: The CoreValve Evolut 34R System is a transcatheter aortic valve implantation system comprised of the following three components:
  1. Evolut 34R Transcatheter Aortic Valve (TAV)
     >
  2. EnVeo R 20Fr Delivery Catheter System (DCS) with EnVeo R InLine Sheath
     >
  3. EnVeo R Loading System (LS)
Period: Enrollment
Arm/Group | CoreValve Evolut R TAVR System 34R Valve
Started | 72
Completed | 60
Not Completed | 12
Not completed — Inclusion Exclusion not met | 9
Not completed — Withdrawal by Subject | 1
Not completed — Expected Enrollment Met | 2
Period: Procedure
Arm/Group | CoreValve Evolut R TAVR System 34R Valve
Started | 60
Completed | 59
Not Completed | 1
Not completed — Death | 1
Period: 1-Month
Arm/Group | CoreValve Evolut R TAVR System 34R Valve
Started | 59
Completed | 54
Not Completed | 5
Not completed — Death | 5
Period: 6-Month
Arm/Group | CoreValve Evolut R TAVR System 34R Valve
Started | 54
Completed | 51
Not Completed | 3
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1
Period: 12-Month
Arm/Group | CoreValve Evolut R TAVR System 34R Valve
Started | 51
Completed | 46
Not Completed | 5
Not completed — Death | 3
Not completed — Withdrawal by Subject | 2
Period: 24-Month
Arm/Group | CoreValve Evolut R TAVR System 34R Valve
Started | 46
Completed | 44
Not Completed | 2
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Period: 36-Month
Arm/Group | CoreValve Evolut R TAVR System 34R Valve
Started | 44
Completed | 35
Not Completed | 9
Not completed — Death | 8
Not completed — Withdrawal by Subject | 1
Period: 48-Month
Arm/Group | CoreValve Evolut R TAVR System 34R Valve
Started | 35
Completed | 27
Not Completed | 8
Not completed — Death | 7
Not completed — Withdrawal by Subject | 1
Period: 60-Month
Arm/Group | CoreValve Evolut R TAVR System 34R Valve
Started | 27
Completed | 24
Not Completed | 3
Not completed — Death | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Groups:
- CoreValve Evolut 34R TAVR System: Treatment of Aortic Stenosis with Medtronic CoreValve Evolut R 34R TAVR System.>
  > CoreValve Evolut 34R TAVR system: The CoreValve Evolut 34R System is a transcatheter aortic valve implantation system comprised of the following three components:>
  1. Evolut 34R Transcatheter Aortic Valve (TAV)>
  2. EnVeo R Delivery Catheter System (DCS) with EnVeo R InLine Sheath>
  3. EnVeo R Loading System (LS)
Arm/Group | CoreValve Evolut 34R TAVR System
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.8 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 58
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With All-cause Mortality
Description: Percentage of participants with all-cause mortality at 30 days
Time Frame: 30 Days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CoreValve Evolut 34R TAVR System
Number analyzed (Participants) | 60
percentage of participants | 1.7 [0.2 to 11.2]

2. Primary Outcome: Percentage of Participants With Stroke (Disabling)
Description: Percentage of participants with disabling stroke (VARC-II definitions) at 30 days
Time Frame: 30 Days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- CoreValve Evolut 34R TAVR System: Treatment of Aortic Stenosis with Medtronic CoreValve Evolut R 34R TAVR System.
  CoreValve Evolut 34R TAVR system: The CoreValve Evolut 34R System is a transcatheter aortic valve implantation system comprised of the following three components:
  1. Evolut 34R Transcatheter Aortic Valve (TAV)
  2. EnVeo R Delivery Catheter System (DCS) with EnVeo R InLine Sheath
  3. EnVeo R Loading System (LS)
Arm/Group | CoreValve Evolut 34R TAVR System
Number analyzed (Participants) | 60
percentage of participants | 0.0 [0.0 to 6.1]

3. Primary Outcome: Device Success Rate
Description: Device Success defined as:
  * Absence of procedural mortality, AND
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location, AND
  * Intended performance of the prosthetic heart valve, defined as the absence of patient prosthesis-mismatch and mean gradient < 20 mmHg (or peak velocity < 3 m/sec), AND
  * Absence of moderate or severe prosthetic valve regurgitation
Time Frame: 24 hours to 7 days post implantation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- CoreValve Evolut 34R TAVR System: Treatment of Aortic Stenosis with Medtronic CoreValve Evolut R 34R TAVR System.
  >
  >
  CoreValve Evolut 34R TAVR system: The CoreValve Evolut 34R System is a transcatheter aortic valve implantation system comprised of the following three components:
  1. Evolut 34R Transcatheter Aortic Valve (TAV)
     >
  2. EnVeo R Delivery Catheter System (DCS) with EnVeo R InLine Sheath
     >
  3. EnVeo R Loading System (LS)
Arm/Group | CoreValve Evolut 34R TAVR System
Number analyzed (Participants) | 60
percentage of participants | 79.2 [65.9 to 89.2]

4. Primary Outcome: The Percentage of Subjects With no More Than Mild Prosthetic Regurgitation at Early Post Procedure Echocardiogram
Description: The percentage of subjects with no more than mild prosthetic regurgitation at early post procedure echocardiogram as assessed by echo core laboratory
Time Frame: 24 hours to 7 days post implantation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CoreValve Evolut 34R TAVR System
Number analyzed (Participants) | 60
percentage of participants | 100.0 [93.9 to 100.0]

5. Secondary Outcome: Percentage of Participants With VARC II Combined Safety Endpoint Event at 30 Days
Description: VARC II composite safety endpoint includes the following components:
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Life-threatening bleeding
  * Acute kidney injury: stage 2 or 3 (including renal replacement therapy).
  * Coronary artery obstruction requiring intervention.
  * Major vascular complication.
  * Valve-related dysfunction requiring repeat procedure (BAV, TAVR, or SAVR)
Time Frame: 30 days post-implantation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CoreValve Evolut 34R TAVR System
Number analyzed (Participants) | 60
percentage of participants | 5.0 [1.6 to 14.7]

6. Secondary Outcome: Percentage of Participants With Life Threatening or Disabling Bleeding
Description: Percentage of participants with life threatening or disabling bleeding - see VARC-2 definitions for classification details
Time Frame: 30 days post-implantation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CoreValve Evolut 34R TAVR System
Number analyzed (Participants) | 60
percentage of participants | 1.7 [0.2 to 11.4]

7. Secondary Outcome: Percentage of Participants With Major Vascular Complication
Description: Percentage of participants with Major vascular complication - see VARC-2 definitions for additional details
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CoreValve Evolut 34R TAVR System
Number analyzed (Participants) | 60
percentage of participants | 1.7 [0.2 to 11.4]

8. Secondary Outcome: Percentage of Participants With Acute Kidney Injury: Stage 2 or 3
Description: Percentage of participants with Acute Kidney Injury: Stage 2 or 3 - see VARC-2 definitions for additional details
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CoreValve Evolut 34R TAVR System
Number analyzed (Participants) | 60
percentage of participants | 0.0 [0.0 to 6.1]

9. Secondary Outcome: Percentage of Participants With Coronary Artery Obstruction
Description: Percentage of participants with coronary artery obstruction - see VARC-2 definitions for additional details
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CoreValve Evolut 34R TAVR System
Number analyzed (Participants) | 60
percentage of participants | 0.0 [0.0 to 6.1]

10. Secondary Outcome: Percentage of Subjects With Valve-related Dysfunction Requiring Repeat Procedure
Description: Percentage of subjects with valve-related dysfunction requiring repeat procedure - see VARC-2 definitions for additional details
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CoreValve Evolut 34R TAVR System
Number analyzed (Participants) | 60
percentage of participants | 0.0 [0.0 to 6.1]

11. Secondary Outcome: Percentage of Subjects With Permanent Pacemaker Implant at 30 Days
Description: Percentage of subjects with new permanent pacemaker implant at 30 days.
Time Frame: 30 days
Population: Subjects with pre-existing pacemaker or internal cardiac defibrillator were excluded from analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CoreValve Evolut 34R TAVR System
Number analyzed (Participants) | 42
percentage of participants | 20.8 [12.1 to 34.3]

12. Secondary Outcome: Percentage of Resheath and Recapture Success
Description: Successful resheathing is defined as Evolut R TAV (including frame) was resheathed into the capsule of the delivery cathether to the desired amount intended, as verified by fluoroscopy.
  Successful recapture is defined as the entire Evolut R TAV (including frame) is resheathed into the capsule of the delivery catheter until there is no gap between the capsule and the tip, as verified by fluoroscopy.
Time Frame: Implant procedure
Population: Success could only be analyzed in subjects where the resheath/recapture feature was used.
Measure: Number; unit: percentage of participants
Arm/Group | CoreValve Evolut 34R TAVR System
Number analyzed (Participants) | 26
percentage of participants | 100.0

13. Secondary Outcome: Hemodynamic Performance Metrics - Mean Gradient
Description: Mean gradient (mmHg) as measured by transthoracic echocardiogram and assessed by echo core laboratory
Time Frame: 30 days
Population: Only participants with echo could be analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CoreValve Evolut 34R TAVR System
Number analyzed (Participants) | 60
mmHg | 6.4 (3.2)

14. Secondary Outcome: Hemodynamic Performance Metrics- Aortic Valve Area
Description: Aortic valve area as measured by transthoracic echocardiogram and assessed by echo core laboratory
Time Frame: 30 Days
Population: Only participants with echo could be analyzed.
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | CoreValve Evolut 34R TAVR System
Number analyzed (Participants) | 60
cm2 | 2.6 (0.7)

15. Secondary Outcome: Hemodynamic Performance Metrics - Total Prosthetic Regurgitation Graded as None/Trace
Description: Total prosthetic regurgitation (none/trace) as measured by transthoracic echocardiogram and assessed by echo core laboratory
Time Frame: 30 days
Population: Only participants with echo could be analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | CoreValve Evolut 34R TAVR System
Number analyzed (Participants) | 58
percentage of participants | 60.3

ADVERSE EVENTS:
Time Frame: All events 6 months, All Cause Mortality 60 months
Groups:
- EVOLUTR 34R: Participants implanted with EVOLUTR 34R device
Arm/Group | EVOLUTR 34R
All-Cause Mortality (participants affected / at risk) | 28/60
Serious Adverse Events (participants affected / at risk) | 34/60
Other Adverse Events (participants affected / at risk) | 48/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EVOLUTR 34R (N=60)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1)
Atrioventricular Block (Cardiac disorders) | 1 (1)
Atrioventricular Block Complete (Cardiac disorders) | 8 (8)
Atrioventricular Block First Degree (Cardiac disorders) | 1 (1)
Bundle Branch Block Left (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 2 (2)
Cardiac Failure Acute (Cardiac disorders) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 2 (3)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 1 (1)
Conduction Disorder (Cardiac disorders) | 1 (1)
Nodal Rhythm (Cardiac disorders) | 1 (1)
Pulseless Electrical Activity (Cardiac disorders) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 2 (2)
Vision Blurred (Eye disorders) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Chest Pain (General disorders) | 2 (2)
Device Embolisation (General disorders) | 1 (1)
Generalised Oedema (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 4 (4)
Sepsis (Infections and infestations) | 1 (1)
Viral Infection (Infections and infestations) | 1 (1)
Arterial Injury (Injury, poisoning and procedural complications) | 1 (1)
Compression Fracture (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Hypoxic-Ischaemic Encephalopathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1)
Confusional State (Psychiatric disorders) | 1 (1)
Glomerulonephritis Membranous (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 4 (4)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 3 (3)
Femoral Artery Dissection (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Peripheral Ischaemia (Vascular disorders) | 1 (1)
All-Cause Mortality (General disorders) | 28 (28)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EVOLUTR 34R (N=60)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Leukocytosis (Blood and lymphatic system disorders) | 8 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 15 (15)
Atrial Fibrillation (Cardiac disorders) | 6 (6)
Atrioventricular Block First Degree (Cardiac disorders) | 12 (13)
Bundle Branch Block Left (Cardiac disorders) | 17 (17)
Extrasystoles (Cardiac disorders) | 4 (4)
Sinus Bradycardia (Cardiac disorders) | 4 (4)
Urinary Tract Infection (Infections and infestations) | 6 (6)
Myocardial Necrosis Marker Increased (Investigations) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5)
Hypervolaemia (Metabolism and nutrition disorders) | 12 (12)
Haematuria (Renal and urinary disorders) | 5 (5)
Renal Failure (Renal and urinary disorders) | 4 (4)
Urinary Retention (Renal and urinary disorders) | 4 (4)
Hypertension (Vascular disorders) | 6 (6)
Hypotension (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No